CLINICAL TRIAL: NCT01471795
Title: The Epidemiology of Ventricular Assist Device-Related Infections
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 08-1093 HP; 5P50HL077096 (NIH)
Record Dates: First submitted 2011-11-07; First posted 2011-11-16 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Study Population: 150 subjects with end-stage heart failure who have been scheduled to undergo device implantation with a VAD, either as a bridge to cardiac transplantation or for destination therapy.

SUMMARY:
Infections often occur after ventricular assist devices (VADs) are placed. These infections can be very serious. The goal of this study is to understand why these infections occur. Bacteria (germs) normally live on our skin and in our noses. After surgery, they can infect the VAD. The investigators will collect cultures of your skin and nose before and after surgery. The investigators will compare these bacteria to bacteria that cause infections. Their genes will be compared to see which ones help the bacteria cause infection.

DETAILED DESCRIPTION:
Infections are one of the most serious of ventricular assist device (VAD) related complications. Many of these infections are associated with significant patient morbidity and mortality. Diagnosis of these infections is often difficult due to the complicated nature of the patient's medical problems, the need for rapid institution of empiric antibiotic therapy and the lack of established criteria that define infection. Staphylococci are among the most common causes of VAD infections. The basis for this high incidence is not well understood but is believed to be in part due to inoculation of staphylococcal commensal flora into wound sites at the time of surgery or thereafter. The goals of this observational study are to develop a better understanding of the pathogenesis and epidemiology of Staphylococcus aureus and epidermidis-VAD infections as well as to develop a set of criteria that can be used to help diagnose the presence or absence of a VAD related infection.

This is a prospective, multi-center, observational study to identify risk factors associated with the development of VAD-related infections. Patients will be followed for up to one year following VAD implantation, time of death or transplantation, whichever comes first. There will be no randomization for this observational study.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years.
2. Approved by the institution's heart failure/transplant committee for VAD implantation, either as a bridge to cardiac transplantation or for destination therapy for end-stage heart failure.
3. Signed informed consent, release of medical information, and HIPAA forms.
4. Expectation of compliance with protocol procedures and study visit schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end-stage heart failure who demonstrate the need for intermediate or long-term support with a VAD.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
The incidence of suspected infections, characterized by infecting organism and location. | Duration of the study, up to one year following VAD implantation, time of death or transplantation, whichever comes first.
  The primary goal is to collect information that describes infections in patients receiving LVADs.

SECONDARY OUTCOMES:
Collect and quantify culture results for suspected infections and the secondary manifestations of infection | Duration of the study, up to one year following VAD implantation, time of death or transplantation, whichever comes first.
  Bacteria normally live on our skin and in our noses.After surgery, they can infect the VAD. We will collect cultures before and after surgery and compare these bacteria to bacteria that cause infections.Their genes will be compared to see which ones help the bacteria cause infection. We hope this will help develop new ways to help prevent VAD infections.
Develop Guidelines to properly diagnose VAD infections | Up to one year following VAD implantation, time of death or transplantation, whichever comes first.
  Information will be collected on patient's medical condition after surgery including blood tests to help determine if an infection is present.
Costs (direct) | Duration of the study, up to one year following VAD implantation, time of death or transplantation, whichever comes first.
  The value of all resources that are consumed in the provision of an intervention or dealing with the side-effects or other current and future consequences linked to it.
Adverse Events | Duration of the study, up to one year following VAD implantation, time of death or transplantation, whichever comes first.
  Since this is an observational study there will be no adverse events directly attributable to a study intervention. However, adverse events that might potentially contribute to the risk or course of VAD-related infections will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Desvigne-Nickens, Study Director — National Heart, Lung, and Blood Institute (NHLBI); Yoshifumi Naka, MD, Study Chair — Columbia University; Michael Parides, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (13):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Sharp Memorial Hospital, San Diego, California
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Jewish Hospital, Louisville, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia Presbyterian Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - LDS Hospital, Salt Lake City, Utah
  - Sacred Heart Medical Center, Spokane, Washington
  - University of Wisconsin Hospital, Madison, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Gordon RJ, Weinberg AD, Pagani FD, Slaughter MS, Pappas PS, Naka Y, Goldstein DJ, Dembitsky WP, Giacalone JC, Ferrante J, Ascheim DD, Moskowitz AJ, Rose EA, Gelijns AC, Lowy FD; Ventricular Assist Device Infection Study Group. Prospective, multicenter study of ventricular assist device infections. Circulation. 2013 Feb 12;127(6):691-702. doi: 10.1161/CIRCULATIONAHA.112.128132. Epub 2013 Jan 11. PMID 23315371
- [Derived] Gordon RJ, Miragaia M, Weinberg AD, Lee CJ, Rolo J, Giacalone JC, Slaughter MS, Pappas P, Naka Y, Tector AJ, de Lencastre H, Lowy FD. Staphylococcus epidermidis colonization is highly clonal across US cardiac centers. J Infect Dis. 2012 May 1;205(9):1391-8. doi: 10.1093/infdis/jis218. Epub 2012 Mar 29. PMID 22457291